CLINICAL TRIAL: NCT01532726
Title: A Non-Interventional, Prospective Study to Assess Seizure Control and Tolerability of Eslicarbazepine Acetate as Adjunctive Therapy to One Baseline Antiepileptic Drug, in Adults With Partial-Onset Seizures With or Without Secondary Generalization
Brief Title: Eslicarbazepine Acetate as Add-On Treatment to One Baseline Antiepileptic Drug (ESLADOBA)
Status: Completed | Type: Observational
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIA-2093-403
Record Dates: First submitted 2012-02-10; First posted 2012-02-14 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Epilepsy
Keywords: Partial-Onset Seizures; Eslicarbazepine Acetate; ESL; BIA 2-093; BIAL
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eslicarbazepine Acetate (ESL): ESL and concomitant medication should be managed by the neurologist according to the respective SPC.Summary of Product Characteristics
  Interventions: Drug: ESL

INTERVENTIONS:
Drug: ESL — ESL 400/800/1200 mg tablets once daily
  Other Names: Zebinix

SUMMARY:
This is a multicenter, non-interventional, prospective study. The observation period comprises at least 6 months, from the initiation of ESL add-on therapy in adult patients with partial-onset epilepsy not sufficiently controlled with one AED, until the first visit that occurs between 6 and 9 months of follow-up. The observation period will end after 9 months of follow-up even if the final assessment is not performed.

DETAILED DESCRIPTION:
To ensure non-interventional status, the neurologist's decision that it is in the patient's best interest to be prescribed with adjunctive ESL has to be made before and independently of his/her decision to include the patient in the study. At all circumstances during the study the patients will be treated and followed according to routine clinical practice. ESL and concomitant medication should be managed by the neurologist according to the respective Summary of Product Characteristics (SPC).In order to reflect real-life practice and to ensure the observational nature of this study, no fixed time-points for study assessment were defined. Intermediate follow-up data will be collected whenever a patient attends to the study's neurologist consultation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient, 18 years or older;
* The patient has an established diagnosis of epilepsy and has experienced at least one partial-onset seizure, with or without secondary generalization, within four weeks prior to initiation of adjunctive ESL;
* The patient is not sufficiently controlled on a current antiepileptic monotherapy and, in the neurologist clinical judgment, it is in the patient's best interest to be prescribed with adjunctive ESL;
* The neurologist's decision to prescribe ESL has been made before and independently of his/her decision to include the patient in this study;
* The patient's treatment is in accordance with the SPC of ESL;
* Written informed consent from the patient (or legally acceptable representative, if the subject is unable to provide informed consent).

Exclusion Criteria:

* Known hypersensitivity to the active substance, carboxamide derivatives (e.g. oxcarbazepine or carbamazepine) or to any of its excipients;
* Patient with 2nd or 3rd degree atrioventricular block;
* Patient treated with an experimental drug within four weeks prior to the introduction of ESL;
* Female patient who is pregnant, lactating, or who is planning to become pregnant during the study period;
* Patient starting ESL outside the approved SPC at enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Partial-Onset Seizures With or Without Secondary Generalization
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
ESL retention rate | 9 months
  Proportion of patients on ESL treatment at the final assessment

SECONDARY OUTCOMES:
CGI-C score at the final assessment. | 9 monthss
  Assessment of effectivenes
Changes in CGI-S score from baseline to final assessment | 9 months
  Assessment of effectivenes
CGI-Efficacy Index scores at the final assessment | 9 months
  Assessment of effectivenes
Proportion of patients who are responders to ESL (at least 50% reduction in seizure frequency) at the final assessment | 9 months
  Assessment of effectivenes
Proportion of seizure-free patients within the 12 weeks prior to final assessment | 9 months
  Assessment of effectivenes
Proportion of seizure-free patients within the 4 weeks prior to final assessment | 9 months
  Assessment of effectivenes
Changes in seizure frequency for partial seizures with or without secondary generalization, from baseline to final assessment | 9 months
  Assessment of effectivenes
Changes in seizure frequency for partial seizures without secondary generalization, from baseline to final assessment | 9 months
  Assessment of effectivenes
Changes in seizure frequency for partial seizures with secondary generalization, from baseline to final assessment | 9 months
  Assessment of effectivenes
Changes in QOLIE-10-P scores from baseline to final assessment | 9 months
  assessment of Quality of life
Occurrence of AEs during the study (overall and treatment-related) | 9 months
  assessment of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: João Chaves, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Hospital Fernando da Fonseca, Lisbon, Lisbon District, Portugal